CLINICAL TRIAL: NCT00606034
Title: A Prospective Trial of U500 Regular Insulin by Continuous Subcutaneous Insulin Infusion in Patients With Type 2 Diabetes and Severe Insulin Resistance Who Have Failed Previous Insulin Regimens
Brief Title: U-500R Insulin In Type 2 Diabetes With Severe Insulin Resistance Via Omnipod
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mountain Diabetes and Endocrine Center (Other)
Responsible Party: Principal Investigator, Wendy Lane MD, Director of Research, Principal Investigator, Mountain Diabetes and Endocrine Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U-500R; U500; B5K-US-X009
Record Dates: First submitted 2008-01-19; First posted 2008-02-01 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes; Insulin Resistance
Keywords: Type 2 diabetes; Insulin Resistance; Continuous Subcutaneous Insulin Infusion; U-500 Insulin; Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects active (Experimental): All subjects will receive the experimental treatment (U-500 insulin via Omnipod) since they have already failed all other previous insulin treatment regimens.
  Interventions: Drug: U-500 Insulin delivered by Omnipod (disposable insulin pump)

INTERVENTIONS:
Drug: U-500 Insulin delivered by Omnipod (disposable insulin pump) — U-500 insulin (concentrated insulin) will be infused continuously subcutaneously using a disposable insulin pump called an Omnipod; the insulin infusion dosage will be individualized to each subject's needs

SUMMARY:
Patients with Type 2 diabetes and severe insulin resistance with very large insulin requirements who have failed all previous insulin regimens using non-concentrated forms of insulin (U100 insulin formulations) will receive 5X concentrated insulin (U500 regular insulin)infused via insulin pump.

DETAILED DESCRIPTION:
Patients with Type 2 diabetes who have severe insulin resistance and very large insulin requirements (over 1.4 units of insulin /kg/day) often fail insulin regimens with persistent poor blood glucose control when standard U-100 insulin formulations are used. This is due in part to poor absorption of the large insulin volumes required using these less concentrated standard insulin preparations. The hypothesis that using a concentrated form of insulin called U-500 Regular insulin and delivering it by infusion via insulin pump will lower the volume of insulin required and therefore improve insulin absorption, which will lead to improved blood glucose control, will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes on stable insulin regimen with or without oral agents for at least 3 months
* HbA1c > 7%
* No significant cardiovascular, renal or other serious medical diseases

Exclusion Criteria:

* HbA1c < 7%
* Chronic renal, hepatic, cardiovascular, or other serious medical illness
* Females of childbearing age not using adequate contraception
* Use of GLP mimetic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy S Lane, MD, Principal Investigator — Mountain Diabetes and Endocrine Center
Locations (1):
- Mountain Diabetes and Endocrine Center, Asheville, North Carolina, United States

REFERENCES:
- [Background] Lane WS. Use of U-500 regular insulin by continuous subcutaneous insulin infusion in patients with type 2 diabetes and severe insulin resistance. Endocr Pract. 2006 May-Jun;12(3):251-6. doi: 10.4158/EP.12.3.251. PMID 16772195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited between Dec 2008 and Dec 2009 from clinic at Mountain Diabetes and Endocrine Center.
Pre-assignment Details: Patients who had failed any previous insulin regimen with HbA1c over 7% and requiring over 100 units of insulin per day were enrolled and switched to treatment with U500 insulin via Omnipod.
Period: Overall Study
Arm/Group | All Subjects Active
Started | 21
Completed | 20
Not Completed | 1
Not completed — incarceration | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects Active
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.86 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Glycemic Control as Assessed by Change in Hemoglobin A1c (HbA1c)
Description: HbA1c is expressed as a percentage. This measurement represents an average of plasma glucose concentration for about 3 months. We will report the change in HbA1c measured at 12 months vs Baseline.
Time Frame: 1 year
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: HbA1c percentage
Groups:
- All Subjects Using U-500 Regular Insulin Via Omnipod: All subjects will receive the experimental treatment (U-500 insulin via Omnipod) since they have already failed all other previous insulin treatment regimens.
Arm/Group | All Subjects Using U-500 Regular Insulin Via Omnipod
Number analyzed (Participants) | 21
HbA1c percentage | -1.23 (1.03)

2. Secondary Outcome: Percentage of Time Spent in Hypoglycemia
Description: For the purposed of this study, hypoglycemia is defined as a blood glucose measurement of less than 70 mg/dl. As part of of this study, subjects will wear a Continuous Glucose Monitor (CGM) for 72 hours to assess glycemic control. The percent of time in hypoglycemia is a part of the download from the CGM.
Time Frame: baseline versus 12 months
Population: ITT (LOCF for 1 subject)
Measure: Mean (Standard Deviation); unit: percent of time spent in hypoglycemia
Arm/Group | All Subjects
Number analyzed (Participants) | 21
percent of time spent in hypoglycemia | -3.7 (4.8)

3. Secondary Outcome: Patient Satisfaction With Insulin Delivery Method Via Insulin Delivery Rating System Questionnaire (IDRSQ)
Description: Overall satisfaction rated on a scale of 0-100 percent with higher numbers indicating greater satisfaction with the insulin delivery method.
Time Frame: Baseline versus 1 year
Population: per protocol
Measure: Mean (Standard Deviation); unit: percent satisfaction
Groups:
- All Subjects: All subjects will receive the IDRSQ at baseline and at Week 52
Arm/Group | All Subjects
Number analyzed (Participants) | 21
percent satisfaction | 90.68 (8.13)

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Subjects will be assessed for adverse events at each study visit and will report serious adverse events via the 24 hour contact number.
Arm/Group | All Subjects Active
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Active (N=21)
Hypoglycemia (Endocrine disorders) | 1 (1) — 1 subject experienced a hypoglycemic event of 39mg/dl which required emergency assistance. The outcome of the event is recovered

LIMITATIONS AND CAVEATS:
Small sample size. Also an uncontrolled pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No